CLINICAL TRIAL: NCT06084260
Title: Comparison of Nutritional Counseling Based on Self-compassion Vs. Diet Approach on Body Dissatisfaction, Food Restriction, and Disordered Eating in Adult Women
Brief Title: Nutritional Counseling Based on Self-compassion Vs. Diet Approach on Body Dissatisfaction and Disordered Eating
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-0634
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Body Dissatisfaction; Disordered Eating
Keywords: body image; eating behaviour; diet; self-compassion
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-compassion group (Active Comparator): Group meetings using a self-compassion approach related to body dissatisfaction and eating issues.
  Interventions: Behavioral: Self-compassion group
- Diet group (Active Comparator): Group meetings using a restricted diet approach related to body dissatisfaction and eating issues.
  Interventions: Dietary Supplement: Diet group

INTERVENTIONS:
Dietary Supplement: Diet group — Individual diet, with caloric restriction, associated with weekly meetings about eating habits modifications.
  Arms: Diet group
Behavioral: Self-compassion group — Weekly meetings using self-compassion techniques to improve body dissatisfaction and eating behavior.
  Arms: Self-compassion group

SUMMARY:
Current evidence has shown that the accepted standard of beauty, where women must be skinny, has increased body dissatisfaction and disordered eating. In order to deal with body dissatisfaction, the practice of restrictive diets - called the diet approach - becomes very often, although it can reinforce disordered eating and has questionable effects on body dissatisfaction. Self-compassion is an approach that proposes a kind and gentle look at body image issues and eating problems, which can be an alternative tool to deal with them. So, this study aims to compare a nutritional approach based on self-compassion techniques x a diet approach on dissatisfaction with body image, food restriction, and disordered eating in women who feel dissatisfied with their bodies.

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted with adult women randomly allocated into two groups - self-compassion (n=38) or diet approach (n=38) - that will follow over eight weeks. Each group will have weekly meetings of 1 hour, working on different subjects related to self-compassion or dietary choices each week, according to each group. The study outcomes are body dissatisfaction, disordered eating, and self-compassion levels, measured through validated questionnaires. Data will be analyzed using Statistical Package for Social Science for Windows software, and differences between the two groups will be evaluated by the Student's T-test or the Mann-Whitney U test, according to sample distribution. The Chi-square test will analyze the associations between the type of approach and all measured outcomes. Significant differences will be considered when the P value <0.05. As a result, the investigators expect that self-compassion will improve body dissatisfaction and attenuate disordered eating more than the diet approach.

ELIGIBILITY:
Inclusion Criteria:

* age between 25 and 59 years;
* access to cell phone and communication apps.

Exclusion Criteria:

* diagnosis of depression, mood disorders (anxiety, bipolar, borderline), eating disorders, or a history of suicidal ideation;
* diagnosis of non-communicable diseases such as diabetes, kidney disease, cardiovascular or neurological diseases.

Ages: 25 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Body dissatisfaction | Baseline and after 8 weeks.
  Dissatisfaction with body image will be assessed using the Body Shape Questionnaire.(BSQ) to identify concerns about body shape and self-deprecation related to physical shape.It has 34 questions related to body image, labeled from 1 to 6, with 1-never, 2-rarely, 3-Sometimes, 4-Frequently, 5-Very often, and 6-Always. The result is obtained by adding all the scores. The minimum score obtained is 34 points, and the maximum is 204. A rating below 80 points considers that the individual has no dissatisfaction; between 80 and 110, there is mild dissatisfaction; between 111 and 140, moderate dissatisfaction; and more than 140, severe dissatisfaction.
Disordered eating | Baseline and after 8 weeks.
  Disordered eating will be measured using The three-factor eating questionnaire - R21 (TFEQ-R21), where three dimensions of eating behavior are evaluated: cognitive restriction, uncontrolled eating, and emotional eating. The higher the score obtained, the more dysfunctional the behavior. A rating below 80 points considers that the individual has no dissatisfaction; between 80 and 110, there is mild dissatisfaction; between 111 and 140, moderate; and more than 140, severe dissatisfaction.

SECONDARY OUTCOMES:
Self-compassion | Baseline and after 8 weeks.
  This outcome will be evaluated through the Self-compassion scale, developed to measure self-compassion in three components: self-judgment versus self-kindness, sense of isolation versus common humanity, and overidentification versus mindfulness.The items are grouped into six subscales: Self-kindness (items 5, 12, 19, 23, 26); Self-judgment (items 1, 8, 11, 16, 21); Common Humanity (items 3, 7, 10, 15); Insulation (items 4, 13, 18, 25); Mindfulness (items 9, 14, 17, 22) and Over-identification (items 2, 6, 20, 24). Each item is rated on a 5-point Likert scale (1 = Almost never; 5 = Almost always). The total score is obtained by adding the scores for all 21 items. Higher scores mean more self-compassion.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina G de Souza, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Ramos AB, da Silva VS, Cardoso DV, de Souza CG. Nutritional approach based in self-compassion versus energy-restricted diet approach in body dissatisfaction and disordered eating in adult women: a protocol for randomized clinical trial. PLoS One. 2025 Jun 2;20(5):e0324030. doi: 10.1371/journal.pone.0324030. eCollection 2025. PMID 40455797